CLINICAL TRIAL: NCT02970877
Title: Fecal Microbiota Transplant From Healthy Lean Donors to Morbidly Obese Individuals: Effect on Insulin Resistance and Other Obesity-related Parameters. A Randomized Controlled Trial.
Brief Title: Stool Transplantation for Treatment of Insulin Resistance in Morbidly Obese Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johane Allard (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); MOUNT SINAI HOSPITAL (Other); University of Toronto (Other)
Responsible Party: Sponsor-Investigator, Johane Allard, Gastroenterologist, Senior Researcher, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-5475
Record Dates: First submitted 2016-06-17; First posted 2016-11-22 (Estimated); Results first posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Obesity, Morbid; Insulin Resistance
Keywords: Fecal microbiota transplant; Intestinal microbiome; Mucosa associated microbiome; Appetite; Metabolome; Depression; Anxiety
MeSH Terms: conditions — Obesity, Morbid; Insulin Resistance; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allogenic treatment group (Experimental): Fecal filtrate from 150 g stool from healthy lean donors
  Interventions: Biological: Fecal filtrate from 150 g stool from healthy lean donors
- Autologous control group (Placebo Comparator): Fecal filtrate from 150 g of the recipient's own stool
  Interventions: Biological: Fecal filtrate from 150 g of the recipient's own stool

INTERVENTIONS:
Biological: Fecal filtrate from 150 g stool from healthy lean donors — 150 g stool from healthy lean donors will be diluted in 0.9% normal saline to a total volume of 450 mL. Preparation from frozen stool.
  Other Names: Intestinal microbiota from healthy lean donors
  Arms: Allogenic treatment group
Biological: Fecal filtrate from 150 g of the recipient's own stool — 150 g stool from the recipient will be diluted in 0.9% normal saline to a total volume of 450 mL. Preparation from frozen stool.
  Other Names: Autologous intestinal microbiota
  Arms: Autologous control group

SUMMARY:
More and more people in Canada and around the world are severely (morbidly) obese, and this is associated with a high risk for poor blood sugar control (insulin resistance, IR) and diabetes. Weight loss is often very hard to achieve for morbidly obese patients. Bariatric surgery is a very effective treatment, but it has some risks and is not available to all patients. Therefore, alternative treatments are needed.

The gut bacteria (intestinal microbiome) might play a role for the development of obesity and IR. Several studies in animals have shown that transferring stool from lean mice or humans into obese animals could lead to weight loss and improve IR. One human study has confirmed this. The investigators are therefore examining, whether transfer of stool from healthy lean people into morbidly obese patients with IR will improve blood sugar control, weight, and other obesity related parameters. This will be done in a randomized controlled trial. Effects on mental health and the bacterial in the mouth related to gum disease will also be assessed.

If successful, fecal transfer could be a new alternative treatment approach for morbidly obese patients or those with IR who do not have access to or do not want to undergo bariatric surgery.

DETAILED DESCRIPTION:
The coupled disorders of morbid obesity and type 2 diabetes (T2D) are a major and growing public health problem in Canada. The Public Health Agency of Canada 2011 report, Obesity in Canada, showed that 5.1% and 2.7% of Canadians had obesity class II (body mass index (BMI) 35.0-39.9) and III (BMI >40 kg/m2), respectively. Morbid obesity is associated with not only T2D (up to 42% of morbidly obese patients), but also cardiovascular complications, non-alcoholic fatty liver disease and sleep apnea, and the prevalence of psychiatric disorders, particularly depression and anxiety, is high in this population. As morbid obesity is very difficult to treat, drastic measures are required, and bariatric surgery is often the only viable treatment option. Bariatric surgery is nowadays a frequently performed procedure (about 400 surgeries/year at the University Health Network (UHN)), and there are different techniques, including gastric banding, sleeve gastrectomy, and Roux-en-Y gastric bypass. Of these procedures, the Roux-en-Y gastric bypass surgery has become the gold standard, and it is highly effective in inducing long-term weight loss and improving or even resolving all of the obesity associated comorbidities. However, bariatric surgery is invasive, costly, has a risk of complications, and requires life-long commitment to a restricted diet. Therefore, a significant proportion of patients with morbid obesity is not willing to undergo the procedure, and a small proportion is excluded from the procedure due to other physical or mental health problems.In addition, depending on the health care system, bariatric surgery might not be available to a large proportion of patients. Regarding the growing rates of obesity and morbid obesity world-wide, less expensive and less invasive alternatives to bariatric surgery are urgently needed.

Even though obesity largely results from an imbalance between energy intake and energy expenditure, it has been shown that several factors, including the genetic background can render individuals susceptible to obesity. Most recently, the role of the intestinal microbiome has been under investigation. It has been shown that obese people have an intestinal microbiome and metagenome that is significantly different from lean controls, and this is even true in identical twins discordant for obesity. In addition, patients with T2D have a different intestinal microbiome than controls. Work done in rodents showed that fecal microbiota transplant (FMT) from lean to obese animals (and vice versa) can affect fat mass and parameters of the metabolic syndrome. It is thus possible that FMT may benefit human obesity with related metabolic abnormalities. FMT is becoming standard therapy for patients with refractory Clostridium difficile colitis and may become a treatment option in other gastrointestinal disorders. Only one human study (n=9) investigated FMT from lean subjects to obese patients (~BMI 35 kg/m2) with metabolic syndrome and showed improvement in insulin sensitivity. Taken altogether, these very exciting results led us to hypothesize that that FMT from healthy lean donors could effectively induce metabolic improvement (i.e. insulin resistance (IR)) and weight loss) by distinct microbe-specific mediated mechanisms. The investigators will examine this in a single-center, double-blind, randomized controlled parallel-group trial (RCT).

Furthermore, emerging evidence shows that the intestinal microbiome, through the gut-brain axis, can influence mood disorders. First animal studies suggest that FMT can transfer depression and anxiety and therefore, FMT from healthy individuals may provide some benefits. Therefore, the investigators will also assess, whether FMT influences depression and anxiety, which are highly prevalent in obese patients. Finally, our Canadian Institutes for Health Research (CIHR) Team Grant, which supports this RCT, is also studying the potential relationship between obesity, T2D and the oral microbiome (OM). Considering that microbes present in the saliva are swallowed in significant numbers-about 10^12 oral bacteria per day-and that this may influence the composition of the intestinal microbiome, the investigators are also exploring the potential relationship between oral and intestinal microbiome and their associations with obesity and T2D. Having a FMT protocol gives us the unique opportunity to further assess this potential relationship and determine if FMT may change OM by improving obesity and metabolic parameters. This has not been previously studied in animals or humans.

The aims of this RCT are to assess whether FMT from healthy lean individuals into morbidly obese patients with IR who decline bariatric surgery, leads to 1) improvement in metabolic parameters: IR, BMI, and other obesity related parameters; 2) improvement in mood disorders: depression and anxiety scores; 3) changes in the intestinal microbiome and metabolome. 4) In addition, by assessing the OM through the FMT protocol and by combining these results with the results of our other protocols in a similar patient population going through bariatric surgery, the investigators will explore the relationship between oral/intestinal microbiome and obesity/metabolic parameters. 5) Furthermore, as planned in our CIHR Team Grant, the investigators will use the FMT from the lean donors and transfer into obese mice to assess the effect of FMT on mechanisms related to glucose metabolism. These additional experiments are not part of this protocol but are mentioned briefly, as stool samples and data from the patients and donors participating in the FMT trial will be used for the other studies in our CIHR Team Grant.

Significance. The number of obese patients is growing world-wide. The investigators are examining here a'medical bypass' solutions to treat the 40-50% of obese patients that meet the criteria set by the National Institutes for Health (NIH) for bariatric surgery (12, 36) but decline (13), or the much larger population of obese patients (BMI 30-40 kg/m2) who may not be considered for surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* age 18 years or older
* morbidly obese (BMI >40 kg/m² or BMI >35-40 kg/m² with other severe weight loss responsive comorbidities)
* referred to the Bariatric Clinic at the Toronto Western Hospital for weight loss surgery, but declining or deferring the surgery
* insulin resistance (HOMA-IR value >2.73)

Exclusion Criteria:

* In the 3 months prior to study entry, regular intake of:

  * non-steroidal anti-inflammatory drugs;
  * iron supplements;
  * prebiotics or probiotics from other than food sources;
  * antibiotics; or
  * any experimental drug
* Type 1 or type 2 diabetes
* chronic gastrointestinal diseases
* previous gastrointestinal surgery modifying the anatomy
* smoking
* pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johane P Allard, MD, Principal Investigator — University Health Network, University of Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The current data sharing plans for the current study are unknown and will be made available at a later date

REFERENCES:
- [Background] Vrieze A, Van Nood E, Holleman F, Salojarvi J, Kootte RS, Bartelsman JF, Dallinga-Thie GM, Ackermans MT, Serlie MJ, Oozeer R, Derrien M, Druesne A, Van Hylckama Vlieg JE, Bloks VW, Groen AK, Heilig HG, Zoetendal EG, Stroes ES, de Vos WM, Hoekstra JB, Nieuwdorp M. Transfer of intestinal microbiota from lean donors increases insulin sensitivity in individuals with metabolic syndrome. Gastroenterology. 2012 Oct;143(4):913-6.e7. doi: 10.1053/j.gastro.2012.06.031. Epub 2012 Jun 20. PMID 22728514
- [Background] Kelly CR, Kahn S, Kashyap P, Laine L, Rubin D, Atreja A, Moore T, Wu G. Update on Fecal Microbiota Transplantation 2015: Indications, Methodologies, Mechanisms, and Outlook. Gastroenterology. 2015 Jul;149(1):223-37. doi: 10.1053/j.gastro.2015.05.008. Epub 2015 May 15. PMID 25982290
- [Background] Hamilton MJ, Weingarden AR, Unno T, Khoruts A, Sadowsky MJ. High-throughput DNA sequence analysis reveals stable engraftment of gut microbiota following transplantation of previously frozen fecal bacteria. Gut Microbes. 2013 Mar-Apr;4(2):125-35. doi: 10.4161/gmic.23571. Epub 2013 Jan 18. PMID 23333862

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Allogenic Treatment Group | Autologous Control Group
Started | 15 | 14
Completed | 15 | 13
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Allogenic Treatment Group | Autologous Control Group | Total
Number analyzed (Participants) | 15 | 13 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 13 | 28
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 45.0 [33.0 to 57.0] | 48.0 [42.0 to 56.0] | 46.5 [37.3 to 56.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 3 | 3 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 15 | 13 | 28
HOMA-IR [Median (Inter-Quartile Range); unit: Index] — Measure of insulin resistance. A person with HOMA-IR > 2.73 is consideered to have insulin resistance. The higher the HOMA-IR, the worse the insulin resistance.
  Index | 3.88 [3.55 to 4.67] | 4.92 [3.94 to 6.55] | 4.34 [3.65 to 5.41]

OUTCOME MEASURES:

1. Primary Outcome: Change in Insulin Resistance Compared to Baseline
Description: Looking at the change in Homeostasis model of assessment for insulin resistance (HOMA-IR). HOMA-IR > 2.73 is considered as insulin resistance. The higher HOMA-IR, the worse the insulin resistance. For this measure, we looked at the change in HOMA-IR. Those with more reduction in HOMA-IR experience more improvement in their insulin resistance.
Time Frame: 1 month, 3 month
Measure: Median (Inter-Quartile Range); unit: Index
Arm/Group | Allogenic Treatment Group | Autologous Control Group
Number analyzed (Participants) | 15 | 13
Index
  Baseline to 1 mo | -0.25 [-0.76 to 2.45] | 1.16 [-0.49 to 3.14]
  Baseline to 3 mo | -0.04 [-0.8 to 2.12] | 0.93 [-0.68 to 2.52]

2. Secondary Outcome: Weight
Description: Body weight (kg)
Time Frame: Baseline, 1 mo, 3 mo
Measure: Median (Inter-Quartile Range); unit: Kg
Arm/Group | Allogenic Treatment Group | Autologous Control Group
Number analyzed (Participants) | 15 | 13
Kg
  Baseline | 126.8 [107.2 to 133.5] | 122.8 [119.0 to 138.2]
  1 mo | 123.8 [107.6 to 134.0] | 122.0 [120.4 to 138.0]
  3 mo | 125.8 [107.8 to 138.6] | 126.4 [120.8 to 134.0]

3. Secondary Outcome: Body Mass Index
Description: Weight (kg)/ height (m^2)
Time Frame: Baseline, 1 mo, 3 mo
Measure: Median (Inter-Quartile Range); unit: kg/m^2
Arm/Group | Allogenic Treatment Group | Autologous Control Group
Number analyzed (Participants) | 15 | 13
kg/m^2
  Baseline | 43.0 [39.0 to 46.9] | 45.1 [40.9 to 50.8]
  1 mo | 43.2 [39.15 to 47.67] | 44.8 [41.4 to 52.1]
  3 mo | 42.64 [39.04 to 47.23] | 44.91 [37.95 to 54.00]

4. Secondary Outcome: Appetite Score
Description: Appetite score according to visual analog scale. Scores range from 0 to 10. In hunger, zero means not hungry at all. In prospective consumption, 0 means "don't think they can eat anything at all" and lower score is better. In sweet craving, zero means "they very much would like to eat something sweet", thus, higher score is better.
Time Frame: Baseline, 1 mo, 3 mo
Measure: Median (Inter-Quartile Range); unit: score on a scale of 1 to 10
Arm/Group | Allogenic Treatment Group | Autologous Control Group
Number analyzed (Participants) | 15 | 13
score on a scale of 1 to 10
  Prospective consumption (Baseline) | 7.3 [4.6 to 8.8] | 6.1 [4.5 to 8.3]
  Prospective consumption (1 mo) | 4.9 [2.3 to 5.3] | 3.9 [2.3 to 5.5]
  Hunger (Baseline) | 5.5 [3.1 to 6.5] | 5.5 [2.0 to 6.6]
  Hunger (3 mo) | 3.6 [2.6 to 4.8] | 2.9 [2.1 to 4.2]
  Sweet craving (Baseline) | 2.8 [1.5 to 5.0] | 1.4 [0.5 to 4.6]
  Sweet craving (3 mo) | 6.8 [4.3 to 9.0] | 3.3 [1.6 to 5.0]

5. Secondary Outcome: Quality of Life Questionnaire
Description: RAND 36-Item Health Survey 1.0 (SF-36). It is a 36-item questionnaire that asks questions about physical functioning, bodily pain, emotional well-being, social functioning, energy/fatigue, and general health perceptions, role limitations due to physical health problems, role limitations due to personal or emotional problems. The lowest score is 0 and the highest score is 100. Higher score shows better overall quality of life.
Time Frame: Baseline, 3 mo
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Allogenic Treatment Group | Autologous Control Group
Number analyzed (Participants) | 15 | 13
score on a scale
  Energy/Fatigue (Baseline) | 43 [35 to 60] | 50 [20 to 50]
  Energy/Fatigue (3 mo) | 55 [35 to 65] | 45 [15 to 55]
  Emotional wellbeing (Baseline) | 78 [48 to 80] | 76 [52 to 80]
  Emotional wellbeing (3 mo) | 80 [64 to 88] | 72 [48 to 88]

6. Secondary Outcome: Depression Score
Description: Montgomery-Åsberg Depression Rating Scale (MADRS) is used in assessing severity od depressive episode. The score for each question is combined for the total score which ranges from 0 to 60. Zero means no depressive episode and 60 means severe depression.
Time Frame: Baseline, 3 mo
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Allogenic Treatment Group | Autologous Control Group
Number analyzed (Participants) | 15 | 13
score on a scale
  Baseline | 5 [1 to 14] | 9 [4 to 12]
  3 mo | 0 [0 to 4] | 12 [2 to 19]

7. Secondary Outcome: Anxiety Score
Description: Hamilton Anxiety Rating Scale (Ham-A) is a questionnaire that assesses anxiety. The scale is 0 to 30. 0 means no anxiety present and 30 means severe anxiety.
Time Frame: Baseline, 3 mo
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Allogenic Treatment Group | Autologous Control Group
Number analyzed (Participants) | 15 | 13
score on a scale
  Baseline | 4 [1 to 13] | 7 [4 to 11]
  3 mo | 1 [0 to 7] | 10 [4 to 12]

8. Other Pre Specified Outcome: Hemoglobin A1c
Description: Blood measurement which measures proportion of glycated hemoglobin to total hemoglobin. This measurement assesses the blood glucose control in the last 3 months. Generally, hemoglobin A1c < 0.060 is normal, 0.060 ≤ hemoglobin A1c <0.065 is prediabetic and ≥ 0.065 is diabetic.
Time Frame: Baseline, 1 mo, 3 mo
Measure: Median (Inter-Quartile Range); unit: ratio glycated Hb to total Hb
Arm/Group | Allogenic Treatment Group | Autologous Control Group
Number analyzed (Participants) | 15 | 13
ratio glycated Hb to total Hb
  Baseline | 0.05 [0.05 to 0.06] | 0.05 [0.05 to 0.06]
  1 mo | 0.06 [0.05 to 0.06] | 0.06 [0.05 to 0.06]
  3 mo | 0.06 [0.05 to 0.06] | 0.06 [0.05 to 0.06]

9. Other Pre Specified Outcome: Change in Intestinal Microbiome in Stool, Composition
Description: Measured by metagenomic sequencing. This measurement assesses the change in bacterial relative abundance level (in percentage) in the stool following the treatment. Higher values of beneficial bacteria and lower values of harmful bacteria is better. Thus, it is expected that post-FMT, beneficial bacteria will increase and harmful bacteria decrease.
Time Frame: Baseline, 1 mo, 3 mo
Measure: Mean (Standard Error); unit: change in percentage
Arm/Group | Allogenic Treatment Group | Autologous Control Group
Number analyzed (Participants) | 15 | 13
change in percentage
  Holdemanella biformis (Baseline to 1mo) | -0.000279 (0.000865) | -0.000201 (0.00239)
  Blautia obeum (Baseline to 1mo) | -0.0282 (0.0546) | -0.00560 (0.545)
  Clostridium spiroforme (Baseline to 1mo) | 0.199 (0.116) | -0.584 (0.545)
  Flavonifractor plautii (Baseline to 1mo) | -0.0426 (0.138) | -0.474 (0.101)
  Collinsella massiliensis (Baseline to 1mo) | 1.15 (3.49) | 0.284 (0.903)
  Escherichia coli (Baseline to 1mo) | -0.00262 (0.0189) | -0.00578 (0.0147)
  Lactococcus lactis (Baseline to 1mo) | 0.345 (0.962) | 0.224 (0.0491)
  Bacteroides xylanisolvens (Baseline to 1mo) | 0.00615 (0.0612) | -0.00135 (0.0228)
  Roseburia intestinalis (Baseline to 3mo) | -0.078 (0.720) | 0.0374 (0.183)
  Roseburia hominis (Baseline to 3mo) | -0.0036 (0.0562) | -0.011 (0.0601)
  Eubacterium eligens (Baseline to 3mo) | -0.60 (0.248) | 0.0393 (0.438)
  Alistipes putredinis (Baseline to 3mo) | 0.0237 (0.352) | 0.0235 (0.212)
  Ruthenibacterium lactatiformans (Baseline to 3mo) | -0.15 (0.309) | 0.235 (0.614)
  Blautia hydrogenotrophica (Baseline to 3mo) | 0.00531 (0.104) | 0.0521 (0.169)

10. Other Pre Specified Outcome: Blood Lipid Profile
Description: Blood measurement assessing the levels of lipid parameters such as cholesterol and LDL. Higher values for LDL and cholesterol may mean the person has dyslipidemia
Time Frame: Baseline, 1 mo, 3 mo
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Allogenic Treatment Group | Autologous Control Group
Number analyzed (Participants) | 15 | 13
mmol/L
  Cholesterol (Baseline) | 4.80 [4.06 to 5.54] | 5.64 [4.82 to 5.80]
  Cholesterol (1mo) | 4.16 [4.02 to 4.97] | 5.47 [4.87 to 5.80]
  LDL (Baseline) | 2.87 [2.38 to 3.41] | 3.32 [2.94 to 3.68]
  LDL (1mo) | 2.62 [2.22 to 2.81] | 3.14 [2.90 to 3.46]
  LDL (3mo) | 2.54 [2.31 to 2.94] | 2.97 [2.67 to 3.43]

11. Other Pre Specified Outcome: Change in Food Intake
Description: Total daily energy intake from 3-day food record
Time Frame: Baseline, 1 mo, 3 mo
Measure: Median (Inter-Quartile Range); unit: kcal
Arm/Group | Allogenic Treatment Group | Autologous Control Group
Number analyzed (Participants) | 15 | 13
kcal
  Baseline | 2002 [1664 to 2743] | 1753 [1307 to 2269]
  1 mo | 1674 [1475 to 1913] | 1787 [1310 to 2169]
  3 mo | 2012 [1555 to 2608] | 1998 [1648 to 2268]

12. Other Pre Specified Outcome: Change in Food Intake
Description: Daily fat intake (% of energy) from 3-day food record
Time Frame: Baseline, 1 mo, 3 mo
Measure: Median (Inter-Quartile Range); unit: percentage of total energy intake
Arm/Group | Allogenic Treatment Group | Autologous Control Group
Number analyzed (Participants) | 15 | 13
percentage of total energy intake
  Baseline | 41.6 [38.5 to 48.8] | 46.7 [38.2 to 49.0]
  1 mo | 40.8 [29.4 to 48.8] | 38.8 [34.5 to 42.2]
  3 mo | 39.2 [28.0 to 44.5] | 41.7 [37.4 to 47.7]

13. Other Pre Specified Outcome: Change in Food Intake
Description: Daily carbohydrates intake (amount g/d, energy and % of energy) from 3-day food record
Time Frame: Baseline, 1 mo, 3 mo
Measure: Median (Inter-Quartile Range); unit: percentage of total energy intake
Arm/Group | Allogenic Treatment Group | Autologous Control Group
Number analyzed (Participants) | 15 | 13
percentage of total energy intake
  Baseline | 39.4 [35.1 to 41.7] | 35.6 [32.3 to 41.8]
  1 mo | 39.5 [31.6 to 51.4] | 34.9 [28.0 to 47.6]
  3 mo | 45.3 [32.3 to 59.0] | 40.7 [33.7 to 42.4]

14. Other Pre Specified Outcome: Change in Food Intake
Description: Daily protein intake (amount g/d, energy and % of energy) from 3-day food record
Time Frame: Baseline, 1 mo, 3 mo
Measure: Median (Inter-Quartile Range); unit: percentage of total energy intake
Arm/Group | Allogenic Treatment Group | Autologous Control Group
Number analyzed (Participants) | 15 | 13
percentage of total energy intake
  Baseline | 16.9 [14.8 to 21.3] | 16.1 [13.8 to 21.7]
  1 mo | 18.6 [16.9 to 20.4] | 18.5 [15.7 to 22.7]
  3 mo | 17.7 [14.2 to 23.0] | 18.8 [14.0 to 21.6]

15. Other Pre Specified Outcome: Change in Food Intake
Description: Daily fiber intake (g) from 3-day food record
Time Frame: Baseline, 1 mo, 3 mo
Measure: Median (Inter-Quartile Range); unit: g
Arm/Group | Allogenic Treatment Group | Autologous Control Group
Number analyzed (Participants) | 15 | 13
g
  Baseline | 21 [17 to 24] | 18 [10 to 21]
  1 mo | 19 [17 to 27] | 14 [11 to 29]
  3 mo | 18 [15 to 32] | 18 [13 to 26]

16. Other Pre Specified Outcome: Physical Activity
Description: Activity log, self-completed
Time Frame: Baseline, 1 mo, 3 mo
Measure: Median (Inter-Quartile Range); unit: min/day
Arm/Group | Allogenic Treatment Group | Autologous Control Group
Number analyzed (Participants) | 15 | 13
min/day
  Baseline | 5.0 [3.3 to 9.9] | 5.0 [2.4 to 8.3]
  1 mo | 4.9 [2.9 to 8.3] | 4.9 [2.1 to 8.3]
  3 mo | 4.0 [1.1 to 5.9] | 3 [2.0 to 5.7]

17. Other Pre Specified Outcome: Stool Metabolomics
Description: Metabolites and molecules in the stool sample measured using nuclear magnetic resonance spectroscopy.
Time Frame: Baseline, 1 mo, 3 mo
Measure: Mean (Standard Deviation); unit: umol/g
Arm/Group | Allogenic Treatment Group | Autologous Control Group
Number analyzed (Participants) | 15 | 13
umol/g
  Butenylcarnitine (Baseline) | 0.000128 (0.0000482) | 0.000168 (0.0000690)
  Butenylcarnitine (3 mo) | 0.000174 (0.0000963) | 0.000109 (0.0000359)
  Indole Acetic Acid (Baseline) | 0.00838 (0.0106) | 0.0186 (0.0283)
  Indole Acetic Acid (3 mo) | 0.0131 (0.0142) | 0.00986 (0.0134)
  Phenylacetic acid (Baseline) | 0.672 (0.368) | 0.491 (0.386)
  Phenylacetic acid (3 mo) | 0.434 (0.233) | 0.673 (0.592)

18. Other Pre Specified Outcome: Serum Metabolomics
Description: Nuclear magnetic resonance spectroscopy
Time Frame: Baseline, 1 mo, 3 mo
Measure: Median (Standard Deviation); unit: umol/L
Arm/Group | Allogenic Treatment Group | Autologous Control Group
Number analyzed (Participants) | 15 | 13
umol/L
  Kynurenine (Baseline) | 2.56 (0.688) | 2.51 (0.468)
  Kynurenine (1 mo) | 2.67 (0.519) | 3.20 (1.02)
  Decenoylcarnitine (Baseline) | 0.227 (0.0696) | 0.264 (0.0623)
  Decenoylcarnitine (3 mo) | 0.226 (0.0648) | 0.305 (0.114)
  Isoleucine (Baseline) | 63.3 (13.9) | 61.6 (8.6)
  Isoleucine (3 mo) | 58.8 (9.3) | 69.8 (18.2)
  Leucine (Baseline | 112 (23.6) | 122 (19.5)
  Leucine (3 mo) | 111 (16) | 135 (33)

ADVERSE EVENTS:
Time Frame: Adverse events were collected at 1month and 3months post-FMT.
Arm/Group | Allogenic Treatment Group | Autologous Control Group
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 11/15 | 10/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allogenic Treatment Group (N=15) | Autologous Control Group (N=13)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (4)
Stomach cramp (Gastrointestinal disorders) | 6 (6) | 2 (2)
Blaoting (Gastrointestinal disorders) | 5 (5) | 4 (4)
Passing more gas than usual (Gastrointestinal disorders) | 8 (8) | 5 (5)
Nausea/vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2)
Foul smelling stool (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2)
abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT02970877/Prot_SAP_000.pdf